CLINICAL TRIAL: NCT04739943
Title: Remote Monitoring of Respiratory Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not available to continue study
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 56494
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Chronic Respiratory Disease; Asthma; Copd
Keywords: digital health; mobile monitoring
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be given access to one or more devices or smartphone/tablet applications. They will then be followed with surveys as well as data from chart review to see how use of one or more elements for remote monitoring may affect their quality of life and overall care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mobile Monitoring (Experimental): Participants will be asked to use a smartphone or tablet application for remote monitoring or respiratory health. They will be followed over time with surveys as well as chart review to assess effects of adding these mobile monitoring elements to their standard care.
  Interventions: Behavioral: Mobile Monitoring

INTERVENTIONS:
Behavioral: Mobile Monitoring — Participants use a smartphone app for self monitoring of respiratory symptoms

SUMMARY:
Recently, interest in ways to monitor and care for patients remotely has significantly increased due to concerns for infection control as well as a way to increase access to regular clinic visits that may be limited for socioeconomic and geographic reasons. However, remote care can be limited by a lack of objective data to help guide clinical care. With respect to respiratory disease, caring for patients remotely may be enhanced by the ability of patients to monitor at home such things as vital signs, lung sounds, and lung function by spirometry. Enhanced methods to follow symptoms and track medication compliance may also be beneficial. These enhancements could improve care and quality of life both for persons with acute respiratory illnesses and those with chronic respiratory disease (such as asthma or COPD).

The purpose of this study is to develop and study methods for patients to monitor their respiratory health at home and make that data available to medical providers to improve their care.

ELIGIBILITY:
Inclusion Criteria:

* age 1 month or older with a diagnosis of chronic respiratory disease (ex. asthma, COPD), an acute respiratory illness or a healthy volunteer
* able to consent or assent with parental consent

Exclusion Criteria:

* people who do not consent
* significant cognitive impairment
* non-English speaking

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
PROMIS-10 survey | Up to 2 years
  The PROMIS Global-10 short form consists of 10 items that assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life.
Asthma Control Test (ACT) | Up to 2 years
  Asthma Control Test is a patient self-administered tool for identifying those with poorly controlled asthma.
  Scores are on a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). Sores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chinthrajah, MD, Principal Investigator — Stanford University, Sean N. Parker Center for Allergy and Asthma Research
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No